CLINICAL TRIAL: NCT04574427
Title: INtra-operative Evaluation of a Novel FLUorescENt C-mEt Tracer in Penile and Tongue
Acronym: INFLUENCE
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: N19IFC
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Head and Neck Cancer; Penile Cancer
Keywords: surgery; fluorescent c-met tracer; penile; tongue
MeSH Terms: conditions — Head and Neck Neoplasms; Penile Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study we evaluate the feasibility of intraoperative visualization of penile and tongue tumours using the fluorescent tracer EMI-137.

DETAILED DESCRIPTION:
This is a single-center, non-randomized, prospective interventional pilot study. Feasibility of intraoperatively visualizing tumour (margins) in penile and tongue tumours using EMI-137 will be investigated. Patients, ≥ 18 years of age, with ≥T1 penile or tongue cancer undergoing primary tumour surgery will be included. All patients will receive an intravenous bolus injection of EMI-137 prior to surgery. Main study parameters/endpoints are: Intraoperative visualization of primary penile or tongue tumours using a dedicated clinical fluorescence camera. The in vivo detected fluorescence signal will be correlated to ex vivo measurements and pathological assessment of the ex-cised tissue.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, prior to performing any protocol related procedures.
* Age ≥ 18 years at time of study entry.
* ≥ T1 penile or tongue squamous cell cancer
* Scheduled for surgical primary tumour resection

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study.
* Pregnant woman
* Abstaining from usage of two forms of barrier contraceptive or actively planning pregnancy within 90 days.
* Severe kidney insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tongue cancer scheduled for primary tumour resection OR Patients with penile cancer scheduled for primary tumour resection.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
tumour visualization by means of c-MET targeted fluores-cence imaging | peri-operative
  The feasibility of intraoperative tumour visualization by means of c-MET targeted fluores-cence imaging will be evaluated, and the imaging result will be correlated to the level of c-MET expression determined using standard immunohistochemistry.

SECONDARY OUTCOMES:
Lymph node visualization by means of c-MET targeted fluores-cence imaging | peri-operative
  Detection and visualization of lymph node metastases in penile and tongue tumour patients
Dysplasia or Cis by means of c-MET targeted fluores-cence imaging | Peri-operative
  Identification of dysplasia or carcinoma in situ in penile and tongue tumours.

CONTACTS AND LOCATIONS:
Overall Officials: Baris Karakullukcu, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute / Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands